CLINICAL TRIAL: NCT01910649
Title: A Phase I/II, Open Label, Escalating Dose, Pilot Study to Assess the Effect, Safety, Tolerability and Pharmacokinetics of Multiple Subcutaneous Doses of Drisapersen in Patients With Duchenne Muscular Dystrophy and to Assess the Potential for Intravenous Dosing as an Alternative Route of Administration
Brief Title: A Phase I/II, Open Label, Escalating Dose, Pilot Study to Assess Effect, Safety, Tolerability and PK of Multiple SC Doses of Drisapersen in Patients With Duchenne Muscular Dystrophy and to Assess the Potential for IV Dosing as an Alternative Route of Administration
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Regulatory approval was not obtained for drisapersen, hence BioMarin is stopping the development of all exon skipping oligonucleotides in DMD.
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 114673; 2007-004819-54 (EudraCT Number)
Record Dates: First submitted 2012-08-02; First posted 2013-07-29 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Muscular Dystrophies
Keywords: drisapersen
MeSH Terms: conditions — Muscular Dystrophies | interventions — PRO051

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Drisapersen (Experimental): Extension phase of treatment. Intravenous dosing of drisapersen will be investigated as an alternative route of administration
  Interventions: Drug: Drisapersen

INTERVENTIONS:
Drug: Drisapersen — Subcutaneous and Intravenous
  Other Names: PRO051

SUMMARY:
The purpose of the extension phase of this study is to determine whether Drisapersen is effective in the treatment of boys with Duchenne muscular dystrophy resulting from a mutation thought to be corrected by exon 51 skipping.

ELIGIBILITY:
Inclusion Criteria:

* Boys aged between 5 and 16 years inclusive.
* Duchenne muscular dystrophy resulting from a mutation correctable by treatment with PRO051.
* Not ventilator dependent.
* Life expectancy of at least six months.
* No previous treatment with investigational medicinal treatment within six months prior to the study.
* Willing and able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

* Aberrant RNA splicing and/or aberrant response to PRO051, detected by in vitro PRO051 assay during screening.
* Known presence of dystrophin in 5% of fibers in a pre-study diagnostic muscle biopsy.
* Severe muscle abnormalities defined as increased signal intensity in >50% of the tibialis anterior muscle at MRI.
* FEV1 and/or FVC <60% of predicted.
* Current or history of liver or renal disease.
* Acute illness within 4 weeks prior to treatment (Day 1) which may interfere with the measurements.
* Severe mental retardation which in the opinion of the investigator prohibits participation in this study.
* Severe cardiac myopathy which in the opinion of the investigator prohibits participation in this study.
* Need for mechanical ventilation.
* Creatinine concentration above 1.5 times the upper limit of normal (age corrected).
* Serum ASAT and/or ALAT concentration(s) which suggest hepatic impairment.
* Use of anticoagulants, antithrombotics or antiplatelet agents.
* Subject has donated blood less than 90 days before the start of the study.
* Current or history of drug and/or alcohol abuse.
* Participation in another trial with an investigational product.

Ages: 5 Years to 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2008-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Acute phase: Safety data | 18 weeks
  Summarized per dose group
Acute phase and Continued Treatment Phase : Pharmacokinetics measured by T1/2, Cmax, Ctrough, 7d, tmax, and volume of distribution and clearance | 18 weeks
  Plasma concentration versus time profiles of PRO051 (GSK2402968)
Acute phase and Continued Treatment Phase : Safety as assessed by the collection of adverse events (AEs) | 72 weeks
  Change from baseline and summarized values
Continued Treatment Phase :Safety as assessed by laboratory parameters | 72 weeks
  Change from baseline and summarized values

SECONDARY OUTCOMES:
Acute phase: Production of exon skip 51 messenger Ribonucleic acid (mRNA) | 18 weeks
Acute phase: Presence of dystrophin expression | 18 weeks
Acute phase: Muscle function | 18 weeks
  Timed tests and 6-minutes walk
Acute phase: Muscle strength | 18 weeks
  Quantitative Muscle Testing [QMT]- Cooperative International Neuromuscular Research Group (CINRG) and Manual Muscle Testing [MMT]
Continued Treatment Phase: Exon skip efficiency | 72 weeks
Continued Treatment Phase Dystrophin expression in muscle biopsy | 72 weeks
Continued Treatment Phase: Muscle function | 300 weeks
  Timed tests and 6-minutes walk
Continued Treatment Phase: Muscle strength | 300 weeks
  Handheld myometry and spirometry

CONTACTS AND LOCATIONS:
Overall Officials: N Goemans, Dr., Principal Investigator — UZ Leuven

REFERENCES:
- [Result] Goemans NM, Tulinius M, van den Akker JT, Burm BE, Ekhart PF, Heuvelmans N, Holling T, Janson AA, Platenburg GJ, Sipkens JA, Sitsen JM, Aartsma-Rus A, van Ommen GJ, Buyse G, Darin N, Verschuuren JJ, Campion GV, de Kimpe SJ, van Deutekom JC. Systemic administration of PRO051 in Duchenne's muscular dystrophy. N Engl J Med. 2011 Apr 21;364(16):1513-22. doi: 10.1056/NEJMoa1011367. Epub 2011 Mar 23. PMID 21428760
- [Derived] Goemans NM, Tulinius M, van den Hauwe M, Kroksmark AK, Buyse G, Wilson RJ, van Deutekom JC, de Kimpe SJ, Lourbakos A, Campion G. Long-Term Efficacy, Safety, and Pharmacokinetics of Drisapersen in Duchenne Muscular Dystrophy: Results from an Open-Label Extension Study. PLoS One. 2016 Sep 2;11(9):e0161955. doi: 10.1371/journal.pone.0161955. eCollection 2016. PMID 27588424